CLINICAL TRIAL: NCT05891392
Title: Early Results Of Coronary Artery Reconstruction For Extensive Coronary Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Alaa Mahmoud Ibrahim, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med-23-5-01MD
Record Dates: First submitted 2023-05-28; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Coronary Reconstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation of early outcome obtained from coronary reconstruction with or without endarterectomy in extensive diseased coronary arteries

ELIGIBILITY:
Inclusion Criteria:

* Primary elective CABG patients Patch anastomosis more than 2 cm

Exclusion Criteria:

* Patients with combined valvular procedure. Previous open heart surgery Patients with EF <40%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing CABG with extensive coronary artery disease who need reconstruction
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Free from ischemia | 6 Months
  Good Revascularisation

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt